CLINICAL TRIAL: NCT03449108
Title: Clinical Study to Assess Efficacy and Safety of LN-145/LN-145-S1 (Autologous Centrally Manufactured Tumor Infiltrating Lymphocytes) Across Multiple Tumor Types
Brief Title: LN-145 or LN-145-S1 in Treating Patients With Relapsed or Refractory Ovarian Cancer, Triple Negative Breast Cancer (TNBC), Anaplastic Thyroid Cancer, Osteosarcoma, or Other Bone and Soft Tissue Sarcomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Iovance Biotherapeutics, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0672; NCI-2018-00918 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0672 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Bone Sarcoma; Dedifferentiated Chondrosarcoma; Giant Cell Tumor of Bone; Malignancy in Giant Cell Tumor of Bone; Malignant Solid Neoplasm; Ovarian Carcinosarcoma; Platinum-Resistant Ovarian Carcinoma; Poorly Differentiated Thyroid Gland Carcinoma; Recurrent Osteosarcoma; Recurrent Ovarian Carcinoma; Refractory Osteosarcoma; Soft Tissue Sarcoma; Thyroid Gland Anaplastic Carcinoma; Thyroid Gland Squamous Cell Carcinoma; Undifferentiated High Grade Pleomorphic Sarcoma of Bone; Triple Negative Breast Cancer
MeSH Terms: conditions — Bone Neoplasms; Giant Cell Tumor of Bone; Osteosarcoma; Ovarian Neoplasms; Sarcoma; Thyroid Carcinoma, Anaplastic; Histiocytoma, Malignant Fibrous; Triple Negative Breast Neoplasms | interventions — aldesleukin; Cyclophosphamide; fludarabine; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ICI Ovarian Cancer, Sarcomas, Triple Negative Breast Cancer (LN-145-S1, nivolumab) (Experimental): Ipilimumab will be administered as a single dose prior to tumor resection. Nivolumab will be administered once prior to tumor resection. Patients receive cyclophosphamide IV over 2 hours on days -7 and -6, fludarabine IV over 15-30 minutes daily on days -5 to -1, LN-145-S1 IV over 45 minutes on day 0 and aldesleukin IV over 30 minutes on days 1-4 for up to 6 doses. Within 12 weeks after receiving LN-145-S1, patients receive nivolumab IV over 30 minutes every 4 weeks in the absence of disease progression or unacceptable toxicity. The second dose will be administered prior to TIL administration and dosing will continue every 4 weeks and continued until unacceptable toxicity, progression, or start of another cancer therapy.
  Interventions: Biological: Aldesleukin; Biological: Autologous Tumor Infiltrating Lymphocytes LN-145; Biological: Autologous Tumor Infiltrating Lymphocytes LN-145-S1; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Ipilimumab; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Thyroid Cohort (LN-145) (Experimental): Patients receive cyclophosphamide IV over 2 hours on days -7 and -6, fludarabine IV over 15-30 minutes daily on days -5 to -1, autologous tumor infiltrating lymphocytes LN-145 IV over 45 minutes on day 0 and aldesleukin IV over 30 minutes on days 1-4 for up to 6 doses.
  Interventions: Biological: Aldesleukin; Biological: Autologous Tumor Infiltrating Lymphocytes LN-145; Drug: Cyclophosphamide; Drug: Fludarabine; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Autologous Tumor Infiltrating Lymphocytes LN-145 — Given IV
  Other Names: Autologous TILs LN-145; Autologous Tumor-infiltrating Lymphocytes LN-145; LN-145; LN145
Biological: Autologous Tumor Infiltrating Lymphocytes LN-145-S1 — Given IV
  Other Names: Autologous TILs LN-145-S1; Autologous Tumor-infiltrating Lymphocytes LN-145-S1; LN 145-S1; LN-145-S1; LN145-S1
  Arms: ICI Ovarian Cancer, Sarcomas, Triple Negative Breast Cancer (LN-145-S1, nivolumab)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: ICI Ovarian Cancer, Sarcomas, Triple Negative Breast Cancer (LN-145-S1, nivolumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
  Arms: ICI Ovarian Cancer, Sarcomas, Triple Negative Breast Cancer (LN-145-S1, nivolumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well autologous tumor infiltrating lymphocytes LN-145 (LN-145) or LN-145-S1 works in treating patients with ovarian cancer, triple negative breast cancer (TNBC), anaplastic thyroid cancer, osteosarcoma, or other bone and soft tissue sarcomas that do not respond to treatment (refractory) or that has come back (relapsed).

LN-145 is made by collecting and growing specialized white blood cells (called T-cells) that are collected from the patient's tumor. LN-145-S1 is made using a modified process that chooses a specific portion of the T-cells. The T cells may specifically recognize, target, and kill the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate efficacy using objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 in each cohort.

SECONDARY OBJECTIVES:

I. Determine the disease control rate (DCR) within and across cohorts. II. Determine the duration of response (DOR). III. Determine progression-free survival (PFS) and overall survival (OS). IV. Further characterize the safety profile of adoptive cell therapy with tumor infiltrating lymphocytes (TIL) across multiple tumor types.

EXPLORATORY OBJECTIVES:

I. Establish duration of tumor-infiltrating lymphocyte (TIL) persistence. II. Compare the molecular and immunological features of tumors before and after TIL therapy.

III. Prospectively evaluate the existing immunotherapy response criteria (immune-related [ir]RECIST) as the best response assessment tool for TIL therapy among a diverse group of solid tumors.

IV. To investigate TIL attributes (CD8 percentage [%], CD27 and CD28 expression) and correlation with response to therapy.

V. Assess tumor marker (CA-125) response in patients who produce this tumor marker.

VI. To assess Health-Related Quality of Life (HRQOL).

OUTLINE: Patients are assigned to 1 of 2 cohorts.

THYROID CANCER COHORT: Patients receive cyclophosphamide intravenously (IV) over 2 hours on days -7 and -6, fludarabine IV over 15-30 minutes daily on days -5 to -1, autologous tumor infiltrating lymphocytes LN-145 IV over 45 minutes on day 0 and aldesleukin IV over 30 minutes on days 1-4 for up to 6 doses.

ICI OVARIAN CANCER, OSTEOSARCOMA, Triple Negative Breast Cancer, or OTHER BONE AND SOFT TISSUE SARCOMAS COHORT: Within 2-4 weeks prior to surgery, patients receive a single dose of nivolumab IV over 30 minutes, followed by a single dose of ipilimumab IV over 30 minutes Patients receive cyclophosphamide IV over 2 hours on days -7 and -6, fludarabine IV over 15-30 minutes daily on days -5 to -1, LN-145-S1 IV over 45 minutes on day 0 and aldesleukin IV over 30 minutes on days 1-4 for up to 6 doses. Within 12 weeks after receiving LN-145-S1, patients receive nivolumab IV over 30 minutes every 4 weeks in the absence of disease progression or unacceptable toxicity.

For cohorts treated without immune checkpoint inhibitors, completion of treatment is defined as having received any volume of LN-145/LN-145-S1 infusion followed by at least 1 dose of adjuvant IL-2. For cohorts treated with TIL + ICI, completion of treatment will correspond to the last dose of nivolumab or IL2 (if the subject is deemed unsuitable to receive adjuvant nivolumab). Patients are followed up at 18 weeks, 6, 9, 12, 18 and 24 months, then every 3 months for at least 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 (Subjects aged 16-70 may be enrolled into the osteosarcoma cohort).
* Subjects must be willing and able to provide informed consent. For patients < 18 years of age, their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Subjects must have an area of tumor amenable to excisional biopsy (core biopsies may be allowed as detailed in protocol) for the generation of TIL separate from, and in addition to, a target lesion to be used for response assessment.
* Any prior therapy directed at the malignant tumor, including radiation therapy, chemotherapy, and biologic/targeted agents must be discontinued at least 28 days prior to enrollment for preparing TIL therapy. Palliative therapy may be received during the screening period with principal investigator (PI) approval for lesions that are not expected to be used for TIL generation or as target lesions.
* Absolute neutrophil count (ANC) >= 1000/mm^3 (within 7 days of enrollment).
* Hemoglobin >= 8.0 g/dL (transfusion allowed) (within 7 days of enrollment).
* Platelet count >= 100,000/mm^3 (within 7 days of enrollment).
* Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) and aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) =< 2.5 x the upper limit of normal (ULN)

  * Patients with liver metastases may have liver function tests (LFT) =< 5.0 x ULN (within 7 days of enrollment).
* Calculated creatinine clearance (Cockcroft-Gault) >= 50.0 mL/min (within 7 days of enrollment).
* Total bilirubin =< 1.5 x ULN (within 7 days of enrollment).
* Prothrombin time (PT) & activated partial thromboplastin time (aPTT) =< 1.5 x ULN (correction with vitamin K allowed) unless subject is receiving anticoagulant therapy (which should be managed according to institutional norms prior to and after excisional biopsy) (within 7 days of enrollment)
* Negative serum pregnancy test (female subjects of childbearing potential) (within 7 days of enrollment)
* Subjects must not have a confirmed human immunodeficiency virus (HIV) infection.
* Subjects must have a 12-lead electrocardiogram (EKG) showing no active ischemia and Fridericia's corrected QT interval (QTcF) less than 480 ms.
* Subjects must also have a negative dobutamine stress echocardiogram. If neither of these tests can be performed, subject may complete alternative cardiac evaluation deemed clinically appropriate based on the recommendation of cardiology.
* Subjects of childbearing potential must be willing to practice an approved highly effective method of birth control starting at the time of informed consent and for 1 year after the completion of the lymphodepletion regimen. Approved methods of birth control are as follows:

  * Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring).
  * Intrauterine device (IUD).
  * Tubal ligation or hysterectomy.
  * Subject/partner status post vasectomy.
  * Implantable or injectable contraceptives.
  * Condoms plus spermicide.
* Able to adhere to the study visit schedule and other protocol requirements.
* Pulmonary function tests (spirometry) demonstrating forced expiratory value (FEV) 1 greater than 65% predicted or forced vital capacity (FVC) greater than 65% of predicted.
* Ovarian cancer cohort only: Subjects must have high-grade non-mucinous histology (carcinosarcomas are allowed).
* Ovarian cancer cohort only: Subjects must have failed at least two prior lines of chemotherapy (i.e. frontline adjuvant chemotherapy plus one additional line for recurrent/progressive disease), and have platinum resistant disease.
* TIL-ICI ovarian cancer cohort only: Same as "ovarian cancer" above.
* TIL-ICI ovarian cancer cohort only: Enrolled after activation of protocol version 2.0.
* Osteosarcoma cohort only: Subjects with osteosarcomas must have relapsed or become refractory to conventional therapy and have received a regimen including some combination of high-dose methotrexate, doxorubicin, cisplatin, and/or ifosfamide.
* Other bone and soft tissue sarcomas cohort only: Subjects with dedifferentiated chondrosarcomas, dedifferentiated giant cell tumor of bone, giant cell tumor of bone, undifferentiated pleomorphic sarcoma of bone, or high-grade unclassified sarcomas of bone must have received at least one prior line of therapy unless no standard first-line therapy exists in which case enrollment as initial therapy is allowed.
* Other bone and soft tissue sarcomas cohort only: Subjects with other soft tissue sarcomas who have received at least one line of therapy.
* TIL-ICI sarcoma cohort only: Subjects with osteosarcomas must have relapsed or become refractory to conventional therapy and have received a regimen including some combination of high-dose methotrexate, doxorubicin, cisplatin, and/or ifosfamide.
* TIL-ICI sarcoma cohort only: Subjects with dedifferentiated chondrosarcomas, dedifferentiated giant cell tumor of bone, giant cell tumor of bone, undifferentiated pleomorphic sarcoma of bone, or high-grade unclassified sarcomas of bone must have received at least one prior line of therapy unless no standard first-line therapy exists in which case enrollment as initial therapy is allowed.
* TIL-ICI sarcoma cohort only: Subjects with other soft tissue sarcomas who have received at least one line of therapy.
* TIL-ICI sarcoma cohort only: Enrolled after activation of protocol version 2.0.
* Anaplastic and poorly-differentiated thyroid cancer cohort only: Pathologic findings supporting the clinical impression of anaplastic thyroid carcinoma. Diagnosis may include consistent with, or suggestive of terminology associated with: anaplastic thyroid carcinoma, undifferentiated carcinoma, squamous carcinoma; carcinoma with spindled, giant cell, or epithelial features; poorly differentiated carcinoma.
* Anaplastic and poorly-differentiated thyroid cancer cohort only: Measurable distant metastatic disease by RECIST v1.1.
* Anaplastic and poorly-differentiated thyroid cancer cohort only: Subjects who are planned for surgical resection of their tumor, or subjects who are planned for surgery to stabilize the airway (i.e., tracheostomy). Subjects who have a stable airway at the time of consent are eligible if there is tumor that can be resected for TIL manufacturing.
* Anaplastic and poorly-differentiated thyroid cancer cohort only: Previous external beam radiation to the neck is allowed as long as there is a measurable lesion that can be biopsied (separate from the area of radiated tumor) and at least one other for RECIST response assessment.
* TIL-ICI-TNBC cohort only: Subjects must have a confirmed diagnosis of metastatic triple negative breast cancer (Stage IV or recurrent) histologically confirmed as per the AJCC staging system.
* Subjects must have TNBC, defined from standard pathologic assays as negative for ER and PR (<10% tumor staining) and negative for HER2 (IHC<3, gene copy number not amplified; per ASCO/CAP guidelines).
* Subjects must have had at least 1 and no more than 3 prior lines of systemic anticancer therapy for metastatic disease.
* The resectable lesion must be a minimum of 1.5 cm in diameter.

Exclusion Criteria:

* Active or uncontrolled intercurrent illness, including but not limited to ongoing or active infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system. Principal investigator (PI) or his/her designee shall make the final determination regarding appropriateness of enrollment.
* Patients with active viral hepatitis.
* Patients who have a left ventricular ejection fraction (LVEF) < 45% at screening.
* Patients with a history of prior adoptive cell therapies.
* Persistent prior therapy-related toxicities greater than grade 2 according to Common Toxicity Criteria for Adverse Events (CTCAE) version (v)4.03, except for peripheral neuropathy, alopecia, or vitiligo prior to enrollment.

  * Patients who have had a documented grade 2 or greater diarrhea or colitis due to previous immunotherapy must have been asymptomatic for at least 6 months or had a normal colonoscopy post checkpoint treatment, by visual assessment, prior to enrollment.
  * Patients with immunotherapy-related endocrinopathies (e.g. hypothyroidism or hypopituitarism, who are stable on hormonal substitution) and controlled with hormonal replacement, are allowed.
* Primary immunodeficiency.
* History of organ or hematopoietic stem cell transplant.
* Chronic steroid therapy, however prednisone or its equivalent is allowed at =< 10 mg/day.
* Patients who are pregnant or nursing.
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his/her designee, would prevent adequate informed consent.
* History of clinically significant autoimmune disease including active, known, or suspected autoimmune disease. Subjects with resolved side effects from prior checkpoint inhibitor therapy, vitiligo, psoriasis, type 1 diabetes or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded.
* History of clinically significant chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease, or other chronic lung disease.
* History of a second malignancy (diagnosed in the last 5 years). Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy. For the thyroid cancer cohort, subjects have a higher likelihood of prior cancers. Therefore, for this cohort, history of prior thyroid cancer or other indolent cancers is not considered exclusionary if in the opinion of the treating physician such cancers are indolent or unlikely to affect the overall prognosis based on the active thyroid cancer.
* History of known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to initiation of lymphodepletion.
* Has received a live vaccine within 30 days prior to the initiation of lymphodepletion.
* Patients who have a contraindication to or history of hypersensitivity reaction to any components or excipients of the TIL therapy or the other study drugs: non-myeloablative-lymphodepletion (NMA-LD) (cyclophosphamide, mesna, and fludarabine); IL-2; antibiotics of the aminoglycoside group (i.e., streptomycin, gentamicin); any component of the TIL infusion product formulation including human serum albumin (HSA), IL-2, and dextran-40, nivolumab or ipilimumab.
* Any other condition that in the investigator's judgement would significantly increase the risks of participation.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 3 years
  Assessed by Response Evaluation Criteria in Solid Tumors version 1.1. Estimation will use 80% confidence intervals by the Wilson score method.

SECONDARY OUTCOMES:
Disease control rate | Up to 3 years
Duration of response | Up to 3 years
Progression free survival | Up to 3 years
  Will be summarized using Kaplan-Meier estimates.
Overall survival | Up to 3 years
  Will be summarized using Kaplan-Meier estimates.
Incidence of adverse events of adoptive cell therapy with tumor infiltrating lymphocytes (TIL) across multiple tumor types | Up to 3 years

OTHER OUTCOMES:
Duration of TIL persistence | Up to 3 years
  Determined by T-cell receptor (TCR) sequencing of infused T cells serially isolated following LN-145/LN-145-S1 infusion, or alternatively iRepertoire assessment of messenger ribonucleic acid for the TCRs.
Response as determined by the immune-related response criteria | Up to 3 years
  Pearson correlation coefficient and linear regression, when appropriate, will be used to quantify the relationship between phenotypic attributes (CD8 percentage [%], CD27 and CD28 expression, etc.) and response to therapy.
Immunological phenotype of LN-145 by multichannel flow cytometry | Day 0
  Pearson correlation coefficient and linear regression, when appropriate, will be used to quantify the relationship between phenotypic attributes (CD8 %, CD27 and CD28 expression, etc.) and response to therapy.
Tumor assessment via immunohistochemistry, TCR sequencing, and transcriptional analysis | Baseline up to 3 years
  Paired t-test will be used to examine the molecular and immunological features of tumors before and after TIL therapy.
Health Related Quality of Life | Up to 24 months
  Assessed per the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Jazaeri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org